CLINICAL TRIAL: NCT06787560
Title: Clinical Study on the Safety and Efficacy of CD7 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation for Non-malignant Blood and Immune System Diseases
Brief Title: CD7 CAR-T Cell Sequential Allo-HSCT for Non-malignant Blood and Immune System Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024023
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Bone Marrow Failure Syndrome
Keywords: CAR-T; Allo-HSCT; Immuno Deficiency Disorders
MeSH Terms: conditions — Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T cells（ CD7 chimeric antigen receptor T cells） (Experimental): Patients or donors undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with CTX、Flu、VP-16 before CAR-T cells infusion. CAR-T cells could be transfused after 48 hours of preconditioning.
  Interventions: Biological: CD7 CAR-T cells injection; Procedure: Allo-HSCT

INTERVENTIONS:
Biological: CD7 CAR-T cells injection — Each subject receive CD7 CAR T-cells by intravenous infusion
Procedure: Allo-HSCT — allogeneic hematopoietic stem cell transplantation

SUMMARY:
A Clinical Study on the Safety and Effectiveness of CD7 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation for Non-malignant Blood and Immune System Diseases

DETAILED DESCRIPTION:
This is a single-arm, open-label clinical trial to evaluate the safety and efficacy of CD7 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation for Non-malignant Blood and Immune System Diseases. It is planned to enroll 12-20 participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Non-malignant blood and immune system diseases include: hereditary bone marrow failure, congenital immune deficiency, hemoglobinopathy and other non-malignant blood and immune system diseases,

  1. Confirmed hereditary bone marrow failure syndrome. Including: Fanconi anemia, congenital pure red cell aplastic anemia, congenital dyskeratosis, Scheux-Day syndrome, congenital neutropenia, various bone marrow failure related congenital thrombocytopenia and other unclassified congenital bone marrow exhaustion diseases;
  2. It meets the criteria of clinical manifestation, immune function and gene diagnosis of immune deficiency disease;
  3. Diagnosed with hemoglobinopathy and dependent on blood transfusions; serum ferritin levels are < 3000 μg/L, with cardiac and hepatic iron content indicating moderate or lower iron overload; documentation of iron chelation therapy (including prescriptions or invoices) for at least three months prior to screening is available; no hydroxyurea, ruxolitinib, decitabine, or cytarabine has been administered in the three months preceding enrollment. The spleen size must not extend beyond the umbilical horizontal line or the midline of the abdomen. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is indicated, and suitable donors for related allo-HSCT are available.
* 2. Serum total bilirubin ≤1.5 times the upper limit of normal value, serum Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal value range;
* 3. Echocardiography showed Left ventricular ejection fraction (LVEF) >50%;
* 4. Pulse oxygen saturation ≥92% (non-oxygen state);
* 5. The estimated survival is more than 3 months;
* 6. ECOG score 0-1;
* 7. Abdominal B-ultrasonography and other examinations were performed to evaluate spleen size. Splenectomy should be evaluated before transplantation for patients with giant spleen;
* 8. Women and men who are fertile must consent to the use of appropriate contraception before entering the study, during study participation, and for 6 months after transfusion (the safety of this therapy for the unborn child is not known, with unknown risks);
* 9. Subjects who are willing to participate in the study are able to understand and have the ability to sign informed consent.

Exclusion Criteria:

* 1. People with a history of epilepsy or other central nervous system disorders;
* 2. Epstein-Barr virus (EBV) DNA positive;
* 3. People with a history of prolonged QT interval or serious heart disease;
* 4. People with active hepatitis B or C virus;
* 5. Tuberculosis, AIDS and other major infectious diseases;
* 6. Sepsis, pulmonary infection, intestinal infection and other major organ infection and poor control, and/or hypersensitive C-reactive protein, procalcitonin significantly elevated;
* 7. People who have previously received other clinical studies and gene therapy;
* 8. Any situation that the investigator believes may increase the risk to the subject or interfere with the test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events
Transplant related mortality rate | Up to 100 days after Treatment
  The proportion of patients who died after transplantation to the total number of transplant patients during the same period

SECONDARY OUTCOMES:
Allogeneic hematopoietic stem cell transplant implantation rate | Up to 100 days after Treatment
  The proportion of the number of patients who achieved hematopoietic reconstitution to the total number of allogeneic hematopoietic stem cell transplantation patients in the same period.
Time to neutrophil and platelet engraftment | Up to 30 days after Treatment
  The time for neutrophils and platelets to reach the implantation criteria after stem cell reinfusion
Disease-feesurvival，DFS | Up to 2 years after Treatment
  The proportion of disease-free patients who survived to the total number of patients who transplanted allogeneic hematopoietic stem cells during the same period.
Overall survival, OS | Up to 2 years after Treatment
  After transplantation until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China